CLINICAL TRIAL: NCT04044326
Title: The Safety and Efficacy of Spherical Microwave Ablation for the Treatment of Malignant Liver Tumors Closed to Inferior Vena Cava
Brief Title: The Safety and Efficacy of Spherical Microwave Ablation for the Treatment of Malignant Liver Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Machine cannot provide
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201802047DIPB
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2019-08

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: 消融
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: microwave ablation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- microwave ablation (MWA) (Experimental): 20 patients with liver cancer, considered for local treatment of liver tumors of size measuring <5 cm and without any signs of extra-hepatic metastasis, will be enrolled to be treated with microwave ablation (MWA)
  Interventions: Procedure: The Solero Microwave Ablation

INTERVENTIONS:
Procedure: The Solero Microwave Ablation — The Solero Microwave Ablation system (Angiodynamics Ltd, USA) with a single microwave applicator operating at a 2.45 GHz will be used to perform MWA

SUMMARY:
Liver cancer including primary hepatocellular carcinoma (HCC) and metastatic liver cancers is one the most common malignancies in the world. Over 10000 new cases per year are diagnosed in Taiwan. Several pre-clinical studies have already demonstrated microwave ablation (MWA) is a safe and effective treatment for live cancers. The system (Solero Microwave Tissue Ablation System) with 2.45 GHz microwave generator could create a spherical ablation zone, and has certificated by CE (Conformité Européenne) mark and U.S. Food and Drug Administration (FDA) approval in 2017. However, there are still few experiences in using MWA for tumor ablation in Taiwan. In this study, the researchers will perform MWA for 20 inoperable patients with liver cancers adjacent to inferior vena cava (IVC). The researchers will appraisal the clinical feasibility and advantage of the system by this study.

DETAILED DESCRIPTION:
Liver cancer including primary hepatocellular carcinoma (HCC) and metastatic liver cancers is one the most common malignancies in the world. Over 10000 new cases per year are diagnosed in Taiwan. Despite the many treatment options, the prognosis of HCC remains dismal. More than 8000 people died of this cancer every year in Taiwan. A majority (70% to 85%) of patients present with advanced or unresectable disease. In contrast, small liver cancers can be cured with an appreciable frequency. Five-year disease-free survival exceeding 50% has been reported for surgical resection, and for the inoperable patients who do not have vascular invasion or extrahepatic spread. Radiofrequency ablation (RFA) is recommended as an alternative curative therapy. However, the main drawback of RFA is its limitation to tumor location. The tumors located adjacent to big vessels such as inferior vena cava (IVC), could not be ablated completely sometimes.

Microwave ablation (MWA) can ablate tumor by higher temperature than RFA, so is supposed not to be diminished by adjacent vessels. Several pre-clinical studies have already demonstrated MWA is a safe and effective treatment for live cancers. The system (Solero Microwave Tissue Ablation System) with 2.45 GHz microwave generator could create a spherical ablation zone, and has certificated by CE mark and FDA approval in 2017. However, there are still few experiences in using MWA for tumor ablation in Taiwan. In this study, we will perform MWA for 20 inoperable patients with liver cancers adjacent to IVC in our hospital. The researchers will evaluate the potential side effect and ablate effect of tumors by abdominal CT or MRI, and the researchers will also follow-up this patients for 4 months to evaluate the complete ablation rate and local recurrence rate. We will appraisal the clinical feasibility and advantage of the system by this study.

ELIGIBILITY:
Patients must meet all of the following inclusion criteria to be eligible for this study:

1. The diagnosis of hepatocellular carcinoma (HCC) or metastatic liver cancers with pathologic proven, and the diagnosis of HCC will be made by pathology / cytology or according to the AASLD(2010) diagnostic criteria. In brief, Nodules larger than 1 cm found on ultrasound screening of a cirrhotic liver should be investigated further with either tri-phase multidetector CT scan or dynamic contrast enhanced MRI. If the appearances are typical of HCC (i.e., hypervascular in the arterial phase with washout in the portal venous or delayed phase), the lesion should be treated as HCC. If the findings are not characteristic or the vascular profile is not typical, a second contrast enhanced study with the other imaging modality should be performed, or the lesion should be biopsied. Biopsies of small lesions should be evaluated by expert pathologists. Tissue that is not clearly HCC should be stained with all the available markers including CD34, CK7, glypican 3, HSP-70, and glutamine synthetase to improve diagnostic accuracy.
2. Unsuitable for surgical resection but local ablation is indicated, however, the distance between tumour and inferior vena cava is smaller than 1 cm.
3. Have at least one, but less than or equal to 3 tumors,
4. Each tumor must be ≤ 5 cm in diameter,
5. Child-Pugh class A-B,
6. Eastern Cooperative Oncology Group (ECOG) score of 0-1,
7. American Society of Anaesthesiologists (ASA) score ≤ 3,
8. Adequate bone marrow and liver function (1). Platelet count ≥ 100 K/Μl(2). Total bilirubin ≦ 3 mg/dL(3). ALT and AST < 5 x upper limit of normal (4). PT-INR ≦ 2.0.
9. The disease status is not suitable to receive transarterial chemoembolization or other standard treatment.
10. Prior Informed Consent Form
11. Life expectancy of at least 3 months.

Exclusion criteria

Patients presenting with any of the following will not be enrolled into this study:

1. Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
2. Received treatment with an investigational agent/ procedure within 30 days prior to microwave ablation
3. Patients who cannot tolerate RFA procedure, including the patients have tumors closed to gall bladder, pancreas, liver hilum and main bile ducts
4. Acute infection or inflammation, acute and severe dysfunction of heart, liver and kidney, and the patients with metallic implantation including pacemaker.
5. Known history of HIV infection
6. Concurrent extrahepatic cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
the efficacy of microwave ablation for the treatment of primary or secondary liver cancers: modified RECIST criteria | up to one year
  The primary measure for this will be the evaluation of tumor response according to the modified RECIST criteria by CT or MR imaging performed 1 month after treatment.

SECONDARY OUTCOMES:
safety and local tumor recurrences | within 30 days of treatment
  The safety endpoint will be treatment-related Serious Adverse Events occurring within 30 days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, MDPHD, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan